CLINICAL TRIAL: NCT02486614
Title: The Effect of Regional Citrate Anti-coagulation on the Coagulation System in Critically Ill Patients Receiving Continuous Renal Replacement Therapy for Acute Kidney Injury - an Observational Cohort Study
Brief Title: Effect of Citrate on the Coagulation System in Patients Receiving CRRT
Acronym: Citroco
Status: Completed | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RJ114/N168
Record Dates: First submitted 2015-06-10; First posted 2015-07-01 (Estimated); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Acute Kidney Failure
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: CRRT — citrate based continuous renal replacement therapy

SUMMARY:
The aim of this study is to evaluate the effect of regional citrate anti-coagulation on different pathways of the coagulation system in critically ill patients with acute kidney injury. This will form the basis for future studies where the investigators plan to focus on patients with premature circuit clotting despite optimal post-filtrate ionised calcium parameters.

DETAILED DESCRIPTION:
Purpose of clinical trial:

To evaluate the effect of regional citrate anti-coagulation on different pathways of the coagulation system in critically ill patients with acute kidney injury.

Patient population:

critically ill patients with acute kidney injury requiring citrate-based continuous renal replacement therapy (CRRT)

Primary objective:

Changes from baseline in a number of measures of coagulability (platelet count; Prothrombin Time; Activated Partial Thromboplastin Time ratio; fibrinogen; d-dimers; Thrombin generation assay; Clot lysis; platelet function analysis 100) in both the blood within the patient's systemic circulation and the CRRT circuit over the course of 72 hours of regional anticoagulation with citrate.

Number of Subjects/Patients:

12 patients with complete data.

Trial Design:

Prospective non-interventional study.

Endpoints:

Change from baseline in a number of measures of coagulability.

Main Inclusion Criteria:

Adult intensive care patients undergoing CRRT with citrate regional anti-coagulation for AKI.

ELIGIBILITY:
Inclusion criteria:

* acute kidney injury treated with citrate based continuous renal replacement therapy (CRRT)
* age >18 years.
* expected to require >72 hours of CRRT.

Exclusion criteria:

* Known preexisting clotting tendency
* Known preexisting bleeding tendency
* Disseminated Intravascular Coagulation (DIC)
* Prior transfusion of any blood product in the 24 hours before enrolment
* Active bleeding (ie. needing blood transfusion) at time of enrolment
* Haemoglobin at time of enrolment <75g/L
* Haematocrit at time of enrolment >0.55
* Patient would refuse Red Blood Cell transfusion (for example Jehova's Witness).
* Platelet count at time of enrolment <100x103/µL
* Treatment with any anticoagulant or antiplatelet agent at time of enrolment or within 7 days of enrolment with the exception of heparin or low molecular weight heparin for DVT prophylaxis.
* Intravenous heparin exposure within 4 hours of commencing citrate anticoagulation.
* Malnourished: BMI <18.5kg/m2 or unplanned weight loss >10% actual body weight (ABW) in preceding 6 months or BMI <20kg/m2 and unplanned weight loss >5% ABW in preceding 6 months.
* CRRT prescribed for an indication other than AKI (for example poisoning).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults with acute kidney injury requiring citrate based continuous renal replacement therapy
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Changes of parameters of coagulability during Continuous Renal Replacement Therapy (CRRT) with citrate anticoagulation | 72 hours
  Changes of coagulation parameters (Full Blood Count, prothrombin time, activated partial thromboplastin time ratio, fibrinogen, d-dimer, thrombin generation, clot lysis and platelet function analysis) during citrate-based CRRT

SECONDARY OUTCOMES:
Determination of baseline coagulation status before initiation of citrate-based CRRT | Before initiation of CRRT
  Determination of parameters of coagulation [Full Blood Count (FBC), prothrombin time (PT), activated partial thromboplastin time ratio (APTTr), fibrinogen, D-dimers, antithrombin activity, protein C activity, free Protein S antigen, resistance to activated protein C screening, homocysteine, prothrombin 20210 mutation test, factor VIII level, Von Willebrand factor antigen, Dilute Russell's Viper Venom Time, dilute activated partial thromboplastin time, anticardiolipin antibodies, anti-beta 2 glycoprotein I antibodies, thrombin generation assay, clot lysis, platelet function 1+2, Thrombin-Antithrombin and platelet function analysis] before initiation of citrate-based CRRT

CONTACTS AND LOCATIONS:
Overall Officials: Marlies Ostermann, PhD, Principal Investigator — Guy's & St Thomas' Foundation Hospital
Locations (1):
- Guy's & St Thomas Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fisher R, Moore GW, Mitchell MJ, Dai L, Crichton S, Lumlertgul N, Ostermann M. Effects of regional citrate anticoagulation on thrombin generation, fibrinolysis and platelet function in critically ill patients receiving continuous renal replacement therapy for acute kidney injury: a prospective study. Ann Intensive Care. 2022 Mar 31;12(1):29. doi: 10.1186/s13613-022-01004-w. PMID 35355147
- [Derived] Fisher R, Lei K, Mitchell MJ, Moore GW, Dickie H, Tovey L, Crichton S, Ostermann M. The effect of regional citrate anti-coagulation on the coagulation system in critically ill patients receiving continuous renal replacement therapy for acute kidney injury - an observational cohort study. BMC Nephrol. 2017 Oct 2;18(1):304. doi: 10.1186/s12882-017-0718-z. PMID 28969597